CLINICAL TRIAL: NCT05843617
Title: Comparison of Bioavailability of Liposomal and Traditional Formulation of Vitamin C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AronPharma Sp. z o. o. (Industry)
Collaborators: Medical University of Warsaw (Other); Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 01-AP-VC
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Bioavailability of Vitamin C
Keywords: Ascorbic Acid; Liposomal Vitamin C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Vitamin C (Experimental): Single oral dose of liposomal vitamin C formulation
  Interventions: Dietary Supplement: Liposomal Vitamin C
- Traditional Vitamin C (Active Comparator): Single oral dose of traditional vitamin C formulation
  Interventions: Dietary Supplement: Traditional Vitamin C

INTERVENTIONS:
Dietary Supplement: Liposomal Vitamin C — 1000 mg of ascorbic acid in liposomal formulation
  Arms: Liposomal Vitamin C
Dietary Supplement: Traditional Vitamin C — 1000 mg of ascorbic acid in traditional formulation
  Arms: Traditional Vitamin C

SUMMARY:
The aim of the study was to compare the profiles of vitamin C serum concentration in healthy volunteers after the single oral administration either in a liposomal or traditional formulation.

DETAILED DESCRIPTION:
The randomized, double-blind, cross-over study was conducted under the supervision of physician on a group of 10 healthy subjects. The volunteers received 1g of vitamin C in a traditional formulation (powder in capsules), and after 14 days of a washout period 1 gram of liposomal formulation (powder in capsules). Venous blood was collected from each participant of the study immediately before the administration of a studied substance and 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 24 hours post the administration.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-65 years old.
* Signed informed consent.
* No injuries or hospitalizations within the last 3 months.
* Refraining from consuming any vitamin C supplements or foods enriched with vitamin C for a period of 72 hours. Limiting excessive consumption of red peppers, parsley (stalks), Brussels sprouts, broccoli, turnip, tomatoes, cabbage, spinach, watercress, citrus fruits, and citrus juices. Not taking acetylsalicylic acid (aspirin, polopiryna, etopiryna) during the study.
* Participants should fast for at least 8-12 hours prior to the administration of the preparations.

Exclusion Criteria:

* Unwilling to give consent.
* Injuries within the last 3 months.
* Cancer (current or past).
* Renal dysfunction (eGFR < 60 ml/min).
* Gastrointestinal disorders (including use of antacids).
* Tobacco use in any form.
* Pregnancy/breastfeeding.
* Patient after organ transplantation, after a stroke, use of anticoagulants, use of immunosuppressants.
* Female patient receiving hormonal therapy (contraception).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Total amount of ascorbic acid that has been absorbed, defined as AUC | baseline, 30 minutes, 1, 2, 3, 4, 6, 8, 10, 24 hours post the administration
  Comparison of the bioavailability of formulations based on the total amount of ascorbic acid that has been absorbed, defined as AUC (area under the curve)
Maximum concentration of ascorbic acid (Cmax) | baseline, 30 minutes, 1, 2, 3, 4, 6, 8, 10, 24 hours post the administration
  Maximum concentration of ascorbic acid achieved in the blood after administration of both formulations

SECONDARY OUTCOMES:
Concentration of ascorbic acid after 24 hours (C24h) | 24 hours post the administration
  Comparison of the concentration achieved in the blood after 24 hours (C24h) from the administration of both formulations

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No